CLINICAL TRIAL: NCT01069692
Title: A Double-blind, Randomized, Placebo-controlled Multi-center Trial to Compare the Phosphate Lowering Efficacy of Different Doses of SBR759 to Placebo
Brief Title: Placebo Versus SBR759 in Lowering Phosphate in Dialysis Patients
Acronym: SBR759
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSBR759A2304; 2008-006097-15 (EudraCT Number)
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2011-07

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Hemodialysis; Hyperphosphatemia; Hyperphosphatemia patients with chronic kidney disease on 3x/week hemodialysis
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: SBR759A
- Arm 3 (Experimental)
  Interventions: Drug: SBR759A
- Arm 2 (Experimental)
  Interventions: Drug: SBR759A
- arm 4 (Experimental): SBR759A
  Interventions: Drug: SBR759A
- arm 5 (Experimental)
  Interventions: Drug: SBR759A

INTERVENTIONS:
Drug: SBR759A — SBR759A 6g daily
  Arms: Arm 3
Drug: SBR759A — Placebo Comparator 0g daily
  Arms: Arm 1
Drug: SBR759A — SBR759A 3g daily
  Arms: Arm 2
Drug: SBR759A — 9g daily
  Arms: arm 4
Drug: SBR759A — 12g daily
  Arms: arm 5

SUMMARY:
This study will compare placebo to 4 different doses of SBR759 to assess the phosphate lowering efficacy in dialysis patients.

ELIGIBILITY:
Inclusion criteria:

1. Men or women of at least 18 years of age
2. Stable maintenance of hemodialysis 3 times per week for 3 months or greater
3. Controlled serum phosphate if under phosphate-binder therapy
4. Patient must either be on a stable phosphate binder dose and are willing to stop their phosphate binder therapy at the beginning of the study, or not have received any phosphate binder therapy for at least 4 weeks prior to screening

Exclusion criteria:

1. Patients who are on peritoneal dialysis
2. Patients who have a transplant or parathyroidectomy scheduled during the study
3. Clinically significant GI disorder
4. Unstable medical condition other than Chronic Kidney Disease
5. Patient is currently being treated with oral iron
6. History of hemachromatosis, or ferritin > 1000 ng/mL
7. Transferrin saturation > 60%
8. Uncontrolled hyperparathyroidism (iPTH > 84.8 pmol/L) Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the change from baseline in 72-hour serum phosphate levels of 4 different doses of SBR759 versus placebo over 4 weeks of treatment | 6 weeks

SECONDARY OUTCOMES:
Evaluate changes in serum phosphate during a 2 week random treatment withdrawal period of SBR759 after 4 weeks treatment | 6 weeks
Evaluate dose-dependent efficacy of SBR759 | 6 weeks
Compare the short-term safety profile and dose-dependent tolerability of SBR759 dosed with meals taken 3 times a day to that of placebo | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Belgium (3):
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Roeselare
- Italy (6):
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Lecco
  - Novartis Investigator Site, Lucca
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Siena

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Fukagawa M, Kasuga H, Joseph D, Sawata H, Junge G, Moore A, Akiba T. Efficacy and safety of SBR759, a novel calcium-free, iron (III)-based phosphate binder, versus placebo in chronic kidney disease stage V Japanese patients on maintenance renal replacement therapy. Clin Exp Nephrol. 2014 Feb;18(1):135-43. doi: 10.1007/s10157-013-0815-7. Epub 2013 May 15. PMID 23670305
- See also: Results for CSBR759A2304 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4647